CLINICAL TRIAL: NCT06455566
Title: Vascular Access for Minimally-invasive Leadless Pacemaker Implantation Through the Right Jugular routE
Acronym: VAMPIRE
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: RYTHMO-2024-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-12 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-02

CONDITIONS: Leadless Pacemaker; Same-day Discharge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Leadless pacemaker implantation through right internal jugular vein
  Interventions: Device: Leadless pacemaker implantation through right internal jugular vein

INTERVENTIONS:
Device: Leadless pacemaker implantation through right internal jugular vein — Leadless pacemaker implantation through right internal jugular vein

SUMMARY:
Leadless pacemakers (LP) are associated with a lower risk of revision compared with transvenous pacemakers. However, LPs implantation is associated with a 0.6% risk of complication at the femoral vein puncture site (e.g. arteriovenous fistula, haemorrhage, pseudoaneurysm, etc.). As a consequence, the need for prolonged in-hospital monitoring after LP implantation though the right femoral (RF)vein is a barrier to same-day discharge. Recently, right internal jugular (RIJ) vein access has emerged an alternative to right RF vein access for LP implantation (with a regulatory approval for MEDTRONIC Micra LP).

The aims of this registry are the following :

* evaluate the feasibility of RIJ access for LP implantation;
* confirm the acute and chronic safety of RIJ access for LP implantation;
* compare RIJ to RF (historical cohort) vein access regarding procedural characteristics and outcomes;
* evaluate the feasibility of same-day discharge avec LP implantation through the RIJ vein.

ELIGIBILITY:
Inclusion Criteria:

* Indication of pacemaker implantation
* Eligible to leadless pacemaker

Exclusion Criteria:

* Contraindication to right internal jugular vein access
* Age < 18 year-old
* Patient already included in a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with a guideline-based pacemaker indication and eligible to leadless pacemaker implantation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Rate of effective of jugular access | [0 - 1 Month]
  Feasibility of jugular access for leadless pacemaker implantation, defined as the percentage of patients with a successful leadless pacemaker implantation through the jugular vein.
Rate of effective same-day discharge | [0 - 1 Month]
  Feasibility of same-day discharge after implantation of a leadless pacemaker through the jugular vein, defined as a successful same-day discharge with no readmission during the first postoperative month.
Incidence of major cardiovascular event | [0 - 12 Month]
  Incidence of major complications related to the implantation of a leadless through the jugular vein:
  * pericardial complications (effusion, tamponade, pericardiocentesis)
  * jugular venous complications (bleeding, hematoma, arteriovenous fistula, vascular surgery)
  * carotid artery complications (bleeding, transient ischemic attack or stroke, vascular surgery)
  * pacemaker malfunction
  * infection
  * cardiac rhythm complications (atrioventricular block, ventricular fibrillation ou tachycardia, cardiac arrest)
  * air embolism

SECONDARY OUTCOMES:
Description of procedural characteristics | During implantation procedure
  Procedural characteristics of leadless pacemaker implantation through the jugular vein (duration, position, number of attempts, ...).

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Angers University Hospital, Angers
  - Caen University Hospital, Caen
  - Grenoble University Hospital, Grenoble
  - Lille University Hospital, Lille
  - Lyon University Hospital, Lyon
  - Metz-Thionville Regional Hospital, Metz
  - Le Millénaire Private Hospital, Montpellier
  - Les Franciscaines Private Hospital, Nîmes
  - Rennes University Hospital, Rennes
  - La Réunion University Hospital, Saint Pierre de La Réunion
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Chami MF, Garweg C, Clementy N, Al-Samadi F, Iacopino S, Martinez-Sande JL, Roberts PR, Tondo C, Johansen JB, Vinolas-Prat X, Cha YM, Grubman E, Bordachar P, Stromberg K, Fagan DH, Piccini JP. Leadless pacemakers at 5-year follow-up: the Micra transcatheter pacing system post-approval registry. Eur Heart J. 2024 Apr 7;45(14):1241-1251. doi: 10.1093/eurheartj/ehae101. PMID 38426911
- [Result] Saleem-Talib S, van Driel VJ, Chaldoupi SM, Nikolic T, van Wessel H, Borleffs CJW, Ramanna H. Leadless pacing: Going for the jugular. Pacing Clin Electrophysiol. 2019 Apr;42(4):395-399. doi: 10.1111/pace.13607. Epub 2019 Feb 25. PMID 30653690
- [Result] Saleem-Talib S, van Driel VJ, Nikolic T, van Wessel H, Louman H, Borleffs CJW, van der Heijden J, Cox M, Ramanna H. The jugular approach for leadless pacing: A novel and safe alternative. Pacing Clin Electrophysiol. 2022 Oct;45(10):1248-1254. doi: 10.1111/pace.14587. Epub 2022 Sep 12. PMID 36031774